CLINICAL TRIAL: NCT05941208
Title: Efficacy of Continuous Fascia Iliaca Block in Hip Surgery in Elderly : a Randomized Controlled Clinical Trial
Brief Title: Efficacy of Continuous Fascia Iliaca Block in Hip Surgery in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Lydia edward aziz zakhary, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Continuous Fascia iliaca block
Record Dates: First submitted 2023-06-24; First posted 2023-07-12 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- study group (Active Comparator): receiving post operative continuous fascia iliaca compartement block for 24 hours
  Interventions: Procedure: continuous fascia iliaca compartment block

INTERVENTIONS:
Procedure: continuous fascia iliaca compartment block — ultrasound Patients were in supine position and the puncture site was selected at 1 cm below the junction point at 1/3 of the connection of anterior superior spine and pubic tubercle. An ultrasound apparatus (Sonosite) high-frequency probe was placed in parallel to the inguinal fold to distinguish the femoral fascia and fascia iliaca, the needle was inserted with out-of-plane technique at an angle of 45° and the tip of the needle was pointed to the head. Once needle-tip placement under the fascia iliaca by hydrolocation was confirmed, the probe was rotated 90° into a longitudinal parasagittal orientation to visualize the needle tip in-plane and to track cephalad spread of the injectate under fascia iliaca, identification of the fascia iliaca plane through the linear probe and introducing epidural catheter 18 G , continuous infusion of bupivacaine 0.25% by a set rate of 7 ml per hour for 24 hours,
  Arms: study group

SUMMARY:
The goal of this clinical trial is to investigate the analgesic effect of ultrasound-guided Continuous fascia iliaca block in very elderly patients with hip fracture after hip surgery compared to systemic analgesia .

The main question[s] it aims to answer are:

* does continuous fascia iliaca block provide adequate post operative analgesia after hip surgery ?
* does it lower the incidence of post operative complications in old age ? Participants will receive continuous fascia iliaca block through ultrasound , introducing epidural catheter 18 G , continuous infusion of bupivacaine 0.25% by a set rate of 7 ml per hour for 24 hours.

Researchers will compare the study group receiving continuous fascia iliaca block to the control group receiving traditional systemic analgesia in the post operative period . to see if the analgesic effect is more effective

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria were randomly assigned into two groups, the control group and the study group, by a computer-generated randomization program. All patients in both group will be informed by the study methods,aim, side effect in clear language, written consent will be taken in clear spoken and written language, All patients of both groups ,once arrived to the OR, monitor will be attached, baseline SBP, DBP,MAP,SPO2,PULSE will be recorded, spinal anesthesia will be performed as follows, after sterilization of the back with bovidon iodine, local anesthesia 3cc of lidocaine 20% will be injected at the level of L3-L4 spine , then injection of 17 mg bupivacaine 0.5% through a 25 spinal needle.

At the end of surgery, Goup 1 will receive continuous fascia iliaca block through ultrasound Patients were in supine position and the puncture site was selected at 1 cm below the junction point at 1/3 of the connection of anterior superior spine and pubic tubercle. An ultrasound apparatus (Sonosite) high-frequency probe was placed in parallel to the inguinal fold to distinguish the femoral fascia and fascia iliaca, the needle was inserted with out-of-plane technique at an angle of 45° and the tip of the needle was pointed to the head.Once needle-tip placement under the fascia iliaca by hydrolocation was confirmed, the probe was rotated 90° into a longitudinal parasagittal orientation to visualize the needle tip in-plane and to track cephalad spread of the injectate under fascia iliaca, identification of the fascia iliaca plane through the linear probe and introducing epidural catheter 18 G , continuous infusion of bupivacaine 0.25% by a set rate of 7 ml per hour for 24 hours The control group will receive traditional analgesia including 50 mg pethidine with a maximum 6 hour interval and 1gm paracetamol as per need .

ELIGIBILITY:
Inclusion Criteria:

* age > 65 years
* American Society of Anesthesiologists (ASA) physical status classification class II,III

Exclusion Criteria:

* age < 65 years
* ASA IIII
* refusal of peripheral nerve block
* infection at the site of injection
* coagulopathy INR > 1.8
* platelets count < 50,000
* known allergy to used medications.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-04-09 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Evaluating the postoperative analgesic effect | 24 hours
  measuring the degree of postoperative analgesia provided by continuous fascia iliaca compartement block using the Visual analogue score for pain ( 11 point scale where 0 indicates no pain, 10 indicates the worst pain imaginable )

CONTACTS AND LOCATIONS:
Overall Officials: Lydia E Zakhary, MD, Principal Investigator — Ainshams U
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

REFERENCES:
- [Background] Rasappan K, Chua ITH, Tey JBL, Ho SWL. The continuous infusion fascia iliaca compartment block: a safe and effective analgesic modality in geriatric hip fracture patients. Arch Orthop Trauma Surg. 2021 Jan;141(1):29-37. doi: 10.1007/s00402-020-03450-2. Epub 2020 May 2. PMID 32361955